CLINICAL TRIAL: NCT03878953
Title: A Phase 3, Open-label Clinical Study of rhPTH(1-84) Treatment in Japanese Subjects With Chronic Hypoparathyroidism
Brief Title: A Clinical Study of rhPTH(1-84) Treatment in Japanese Participants With Chronic Hypoparathyroidism
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP634-301; JapicCTI-194828 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Chronic Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- rhPTH(1-84) (Experimental): Participants will receive a SC injection of initial dose of 50 mcg of rhPTH(1-84) once daily (QD) in the thigh (alternate thigh every day). If albumin-corrected serum calcium (ACSC; [mg/dL] = serum calcium [mg/dL] +0.8*[4-serum albumin (g/dL)]) is >2.25 mmol/L (>9.0 mg/dL), a starting dose of 25 mcg will be considered. At 4 week intervals the rhPTH(1-84) dose may be increased in 25 mcg increments to a maximal dose of 100 mcg SC QD. At any time during the study as needed for safety reasons, rhPTH(1-84) doses may be decreased in 25 mcg decrements to a minimum of 25 mcg QD. If the ACSC is >2.97 mmol/L (>11.9 mg/dL), then the investigational product should be stopped until the calcium level is corrected.
  Interventions: Drug: rhPTH(1-84)

INTERVENTIONS:
Drug: rhPTH(1-84) — Participants will receive a SC injection of initial dose of 50 mcg of rhPTH(1-84) once daily (QD) in the thigh (alternate thigh every day). If albumin-corrected serum calcium (ACSC; [mg/dL] = serum calcium [mg/dL] +0.8*[4-serum albumin (g/dL)]) is >2.25 mmol/L (>9.0 mg/dL), a starting dose of 25 mcg will be considered. At 4 week intervals the rhPTH(1-84) dose may be increased in 25 mcg increments to a maximal dose of 100 mcg SC QD. At any time during the study as needed for safety reasons, rhPTH(1-84) doses may be decreased in 25 mcg decrements to a minimum of 25 mcg QD. If the ACSC is >2.97 mmol/L (>11.9 mg/dL), then the investigational product should be stopped until the calcium level is corrected.

SUMMARY:
This clinical study aims to evaluate the safety and efficacy of repeated dosing of recombinant human parathyroid hormone (rhPTH[1-84]) in Japanese participants with chronic hypoparathyroidism for a 26-week period.

ELIGIBILITY:
Inclusion Criteria:

* The participant has signed and dated the informed consent form.
* The participant is an adult male or female 20 to 85 years of age inclusive.
* The participant is living in Japan and is Japanese; in this case, Japanese is defined as having been born in Japan, with Japanese parents, and Japanese maternal and paternal grandparents.
* The participant has a diagnosis of chronic hypoparathyroidism with an onset of 18 months or more prior to screening. The diagnosis is based on historical biochemical evidence of hypocalcemia in the setting of a concomitant inappropriately low serum intact parathyroid hormone (PTH). If such evidence is not available the diagnosis of chronic hypoparathyroidism must be confirmed by the Shire medical monitor based on other compelling medical history.
* The participant has been treated with active vitamin D therapy with alfacalcidol greater than or equal to (>=) 1 microgram (mcg) per day (or an equivalent dose of calcitriol of >=0.5 mcg per day or falecalcitriol >=0.3 mcg per day) prior to baseline.
* The participant has indicated a willingness and ability to perform daily subcutaneous (SC) self-injections of study medication (or will have a designee, ie, a family member or caregiver, to perform injections).
* Females of childbearing potential must agree to comply with the contraceptive requirements of the protocol.
* The participants who are less than (<) 25 years old demonstrate radiological evidence of epiphyseal closure at screening based on bone age X-ray (single posteroanterior X-ray of the left wrist and hand).
* The participant meets 1 of the following criteria:

  1. If not receiving thyroid hormone replacement therapy, the participant has a serum thyroid stimulating hormone (TSH) level within normal laboratory limits at screening.
  2. If receiving thyroid hormone replacement therapy, the dose must have been stable for at least 3 months prior to screening and serum TSH level within the reference range for the laboratory.
* The participant has a 25-hydroxyvitamin D level >=50 nanomoles per litre (nmol/L) (20 nanogram per milliliter [ng/mL]) and < upper limit of normal (ULN) of the laboratory reference range.
* The participant has a serum creatinine laboratory value of <132.6 micromoles per liter (mcmoles/L) (1.5 milligram per deciliter [mg/dL]).
* The participant has a serum magnesium level within the laboratory reference range at baseline.
* The participant is not adequately controlled with standard therapy within 6 months of screening based upon the opinion of the investigator and approval by the sponsor's medical monitor. For example:

  1. Hypocalcemia (albumin-corrected serum calcium <8.0 mg/dL) or
  2. Hypercalciuria (urine calcium [mg/dL]/creatinine [mg/dL] ratio >0.4 or 24 hour urine calcium excretion >7.5 millimoles (mmol) [300 milligram {mg}]/24 hours in men and >6.25 millimoles (mmol) [250 mg]/24 hours in women) or,
  3. Symptoms of hypoparathyroidism.

Exclusion Criteria:

* The participant and/or legally authorized representative(s) is unable to understand the nature, scope, and possible consequences of the study.
* The participant is unable to comply with the protocol, eg, uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for evaluations, or is otherwise unlikely to complete the study, as determined by the investigator or the medical monitor.
* The participant has any disease that might affect calcium metabolism or calcium-phosphate homeostasis other than hypoparathyroidism, such as active hyperthyroidism, Paget's disease, type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus (hemoglobin A1c [HbA1c] >8%), severe and chronic cardiac, liver or renal disease, Cushing's syndrome, neuromuscular disease, rheumatoid arthritis, myeloma, pancreatitis, malnutrition, rickets, recent prolonged immobility, active malignancy, primary or secondary hyperparathyroidism, a history of parathyroid carcinoma, hypopituitarism, acromegaly, or multiple endocrine neoplasia types I and II.
* The participant has a known history of hypoparathyroidism resulting from an activating mutation in the CaSR gene or impaired responsiveness to PTH (pseudohypoparathyroidism).
* The participant is taking prohibited medications (listed below) or other drugs known to influence calcium and bone metabolism during their respective prohibited periods.

  a) The following prohibited medications should not be taken within the specified number of days prior to the first dose of rhPTH(1-84): i) 30 days: loop diuretics, thiazide diuretics, phosphate binders (other than calcium carbonate), calcitonin, cinacalcet hydrochloride.

ii) 90 days: lithium. iii) 127 days: denosumab. iv) 180 days: digoxin, raloxifene hydrochloride, estrogens and progestins for hormone replacement therapy, methotrexate, systemic corticosteroids, oral bisphosphonates*.

v) 365 days: sodium fluoride, intravenous bisphosphonates*. Note: *The length of the washout period is dependent on the route of administration of bisphosphonate that is being used by the participant.

* The participant has previous treatment or participation in an investigational trial with PTH-like drugs, including PTH(1-84), PTH(1-34) or other N terminal fragments or analogs of PTH or PTH-related protein within 6 months prior to screening.
* The participant has nonhypocalcemic seizure disorder/epilepsy with a history of a seizure within the previous 6 months prior to screening; note that participant with a history of seizures due to hypocalcemia are allowed.
* The participant has any disease or condition, in the opinion of the investigator, which has a high probability of precluding the participant from completing the study or that the participant cannot or will not appropriately comply with study requirements.
* The participant has participated in any other investigational trial in which receipt of investigational drug or device occurred within 6 months prior to screening for this study.
* The participant is pregnant or breastfeeding.
* The participant has a history of diagnosed drug or alcohol dependence within the previous 3 years.
* The participant has a history of gout.
* The participant has disease processes that may adversely affect gastrointestinal absorption, including but not limited to short bowel syndrome, bowel resection, tropical sprue, celiac disease, ulcerative colitis, and Crohn's disease.
* The participant has chronic or severe cardiac disease including, but not limited to, heart failure (according to the New York Heart Association classification Class II to Class IV) (Dolgin and NYHA 1994), arrhythmias, bradycardia (resting pulse rate <50 beats/minute), or hypotension (systolic and diastolic blood pressures <100 and 60 millimeters of mercury (mmHg), respectively).
* The participant has a history of cerebrovascular accident.
* The participant has a known or suspected intolerance or hypersensitivity to the investigational product, PTH derivatives, or any of the stated ingredients.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-31 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Responders at Week 26 | Week 26
  Number of participants who achieved an albumin-corrected total serum calcium concentration that is maintained or normalized compared to baseline and does not exceed the upper limit of the reference range for the laboratory, at least a 50% reduction from baseline amounts of active vitamin D therapy and at least a 50% reduction from the baseline oral calcium supplement dose (this criterion will be considered met if the participant's baseline calcium dose is <1000 mg and it does not increase during the study will be reported.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From start of study treatment up to 30 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this study treatment. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with an investigational product or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the investigational product or medicinal product.

SECONDARY OUTCOMES:
Change From Baseline in Serum Phosphate Level | Baseline, Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 26 and 30
  Change from baseline in serum phosphate level will be reported.
Change From Baseline in Urine Calcium Level | Baseline, Week 26
  Change from baseline in urine calcium level will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- Japan (10):
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - University of Occupational and Environmental Health Japan, Kitakyushu-shi, Fukuoka
  - Osaka City University Hospital, Osaka, Osaka
  - Shimane University Hospital, Izumo-shi, Shimane
  - Tokushima University Hospital, Tokushima, Tokushima
  - University of Tokyo Hospital, Bunkyō City, Tokyo-To
  - The Cancer Institute Hospital of JFCR, Kōtoku, Tokyo-To
  - Toranomon Hospital, Minatoku, Tokyo-To
  - Keio University Hospital, Shinjuku-ku, Tokyo-To
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo-To

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be reidentified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd94db2bf003ab47112